CLINICAL TRIAL: NCT03782480
Title: A Placebo-controlled Study Examining the Morphological/Biochemical Effects of Intrarosa on the Vulvar Vestibule and Vagina in Women With Genitourinary Syndrome of Menopause/Vulvovaginal Atrophy
Brief Title: Examining Effects of Intrarosa in Women With Genitourinary Syndrome of Menopause/Vulvovaginal Atrophy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Vulvovaginal Disorders (Other)
Collaborators: EndoCeutics Inc. (Industry)
Responsible Party: Principal Investigator, Andrew T. Goldstein, MD, Study Principle Investigator, Center for Vulvovaginal Disorders
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGEC-10
Record Dates: First submitted 2018-12-05; First posted 2018-12-20 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Menopause; Genitourinary Syndrome of Menopause; Vulvovaginal Atrophy; Menopause Syndrome; Dyspareunia
MeSH Terms: conditions — Dyspareunia | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrarosa (Active Comparator): Daily intravaginal administration at bedtime of one insert containing 6.5mg (0.50%) prasterone for 26 weeks
  Interventions: Drug: Intrarosa
- Placebo (Placebo Comparator): Daily intravaginal administration at bedtime of one insert containing placebo for 26 weeks
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Intrarosa — Prasterone intravaginal inserts
  Other Names: prasterone; Dehydroepiandrosterone; DHEA
  Arms: Intrarosa
Drug: Placebos — Placebo intravaginal inserts
  Arms: Placebo

SUMMARY:
Tissues of the genitals of women are both androgen (testosterone) and estrogen dependent. The clitoris, vestibule, urethra, anterior vaginal wall, peri-urethral tissue, and pelvic floor all depend on androgens for normal function. In addition, the glands, which secrete lubrication during sexual arousal, also require androgens to function. Deficiencies of both estrogens and androgens occur naturally during menopause. Menopause-related deficiencies of these hormones lead to thinning in the tissues of the genital and urinary systems which have been termed Genitourinary Syndrome of Menopause (GSM). Patients with GSM will frequently complain of dryness and/or pain during sexual intercourse.

Historically, GSM treatment involved both androgens and estrogens, However, over the past few decades estrogen based therapies have become much more common. More recently, clinical trials have demonstrated that local vaginal dehydroepiandrosterone (Intrarosa®) improves symptoms in menopausal women who have moderate to severe pain with intercourse.

Intrarosa® vaginal inserts are a prescription medicine approved by the U.S. Food and Drug Administration (FDA) used in women after menopause to treat moderate to severe pain during sexual intercourse caused by changes in and around the vagina that happen with menopause.

DETAILED DESCRIPTION:
Tissues in the genitourinary system are both androgen- and estrogen-dependent. The clitoris, vestibule, urethra, anterior vaginal wall, peri-urethral tissue, and pelvic floor are androgen-responsive. In addition, the minor vestibular glands and the major vestibular glands (Bartholin's and Skene's) are androgen-dependent, mucin-secreting glands. Deficiencies of both estrogens and androgens can occur both naturally during menopause or iatrogenically because of certain medications (e.g. Depo Lupron, spironolactone) or surgically (oophorectomy). Menopause-related deficiencies of these sex hormones lead to atrophic changes in the genitourinary system which have been termed genitourinary syndrome of menopause (GSM).

While erythema is a nonspecific finding in atrophic tissue, focal painful erythema in the androgen-dependent vestibule, particularly near the ostia of the Bartholin's glands (4:00 and 8:00 o'clock) and Skene's glands (1:00 and 11:00 o'clock) or lesser vestibular glands, is highly suggestive of GSM. Patients with GSM will frequently complain of penetrative dyspareunia and experience allodynia with the cotton swab palpation of the vulvar vestibule. During examination of the vulvar vestibule, the examiner might note general pallor with superimposed erythema. Physical exam can be improved by magnification (i.e. vulvoscopy).

Historically, GSM treatment involved both androgens and estrogens. However, in the absence of information about intracrinology, over the past few decades, estradiol-based therapies have been used exclusively. More recently, double-blind, placebo controlled clinical trials demonstrated that local vaginal dehydroepiandrosterone (Intrarosa®) improves symptoms in postmenopausal women including moderate to severe dyspareunia. These trials have demonstrated improvement in both subjective measures (such as improvement in dyspareunia) as well as objective measurement of vaginal health (improved vaginal maturation index, decreased vaginal pH) but they have not attempted to demonstrate improvement in the health of the vulvar tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women aged 40 to 80 years.
2. Women who have self-identified at screening pain at sexual activity as moderate to severe and most bothersome symptom of vulvovaginal atrophy (Refer to Vaginal Atrophy Symptoms Questionnaire (VASQ-MBS)).
3. Women having ≤5% of superficial cells on vaginal smear at screening.
4. Women having a vaginal pH above 5 at screening.
5. Willing to participate in the study and sign an informed consent.

Exclusion Criteria:

1. Clinically significant metabolic or endocrine disease (including diabetes mellitus) not controlled by medication.
2. Use of estrogen injectable drug therapy and/or progestin implant within 6 months prior to screening visit.
3. Oral estrogen, progestin or DHEA exposure or intrauterine progestin therapy within 8 weeks prior to screening visit.
4. Vaginal hormonal products (rings, creams, gels or tablets) or transdermal estrogen alone or estrogen/progestin products within 8 weeks prior to screening visit.
5. Previous treatment with androgens or anabolic steroids within 3 months prior to screening visit (see Appendix 15.1 - Concomitant medications).
6. Confirmed clinically significant depression (not controlled by standard therapy) or confirmed history of severe psychiatric disturbance.
7. The administration of any investigational drug within 30 days of screening visit.
8. Clinically significant abnormal serum biochemistry, urinalysis or hematology (as per Investigator's assessment who should take into account the patient's pre-baseline conditions).
9. Uterine palpable fibroids.
10. Uterine prolapse (when the cervix reaches labia minora at gynecologic exam).
11. Subjects who suffer from vulvar lichen sclerosus or any vulvar dermatological disorder that affects the vulvar vestibule or vagina.
12. Chronic use of narcotics or alcoholism during the last 5 years.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-02 (Estimated); Primary Completion 2021-01-02 (Estimated); Study Completion 2021-01-02 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in morphological content of vulvar and vaginal cells | 2 years
  Changes from baseline in density of androgen, estrogen and progesterone receptors. Unit of measure to be determined.
Changes from baseline in morphological content of vulvar and vaginal cells | 2 years
  Changes from baseline in tissue steroid concentrations. Unit of measure to be determined.
Changes from baseline in morphological content of vulvar and vaginal cells | 2 years
  Changes from baseline in blood steroid concentration. Unit of measure to be determined.
Changes from baseline in protein content of vulvar and vaginal cells | 2 years
  Changes from baseline in mucin. Unit of measure to be determined.
Changes from baseline in enzymatic content of vulvar and vaginal cells | 2 years
  Changes from baseline in enzymatic content (HSD17B5, HSD3B1, 5alphaRED2, aromatase, HDS17B1, sulfotransferase 2A1, sulfatase and UGT2B). All enzymes have the same unit of measure. Unit of measure to be determined.
Changes from baseline in antigen content of vulvar and vaginal cells | 2 years
  Changes from baseline in PGP9.5. Unit of measure to be determined.
Changes from baseline in antigen content of vulvar and vaginal cells | 2 years
  Changes from baseline in Ki-67 antigen. Unit of measure to be determined.

SECONDARY OUTCOMES:
Mean change from baseline in subject's scores on pain severity subscale VPAQ | 2 years
  The Vulvar Pain Assessment Questionnaire (VPAQ) was developed to assess the dimensions of the pain experience in studies of chronic pain. It consists of 6 primary (pain severity, emotional response, cognitive response, and interference with life, sexual function, and self-stimulation/penetration) and 3 supplementary subscales (pain quality, coping skills, and partner factors). The pain severity subscale of the VPAQ consists of 3 pairs of verbal rating scale that test both pain intensity and pain affect. Each verbal rating scale is a 5-point scale with the following options: none=0, mild=1, moderate=2, severe=3, and worst possible=4. The calculated mean produces the overall score for the pain severity subscale ranging from 0-4 (4 is the worst score).

CONTACTS AND LOCATIONS:
Overall Officials: Fernand Labrie, MD, Study Director — EndoCeutics Inc.
Locations (2):
- United States (2):
  - The Centers for Vulvovaginal Disorders, Washington D.C., District of Columbia
  - The Centers for Vulvovaginal Disorders, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Labrie F, Martel C, Pelletier G. Is vulvovaginal atrophy due to a lack of both estrogens and androgens? Menopause. 2017 Apr;24(4):452-461. doi: 10.1097/GME.0000000000000768. PMID 27875388
- [Background] Kingsberg S, Kellogg S, Krychman M. Treating dyspareunia caused by vaginal atrophy: a review of treatment options using vaginal estrogen therapy. Int J Womens Health. 2010 Aug 9;1:105-11. doi: 10.2147/ijwh.s4872. PMID 21072280
- [Background] Nappi RE, Palacios S. Impact of vulvovaginal atrophy on sexual health and quality of life at postmenopause. Climacteric. 2014 Feb;17(1):3-9. doi: 10.3109/13697137.2013.871696. PMID 24423885
- [Background] Labrie F. Intracrinology. Mol Cell Endocrinol. 1991 Jul;78(3):C113-8. doi: 10.1016/0303-7207(91)90116-a. PMID 1838082
- [Background] Archer DF, Labrie F, Bouchard C, Portman DJ, Koltun W, Cusan L, Labrie C, Cote I, Lavoie L, Martel C, Balser J; VVA Prasterone Group. Treatment of pain at sexual activity (dyspareunia) with intravaginal dehydroepiandrosterone (prasterone). Menopause. 2015 Sep;22(9):950-63. doi: 10.1097/GME.0000000000000428. PMID 25734980
- [Background] Labrie F, Archer DF, Koltun W, Vachon A, Young D, Frenette L, Portman D, Montesino M, Cote I, Parent J, Lavoie L, Beauregard A, Martel C, Vaillancourt M, Balser J, Moyneur E; VVA Prasterone Research Group. Efficacy of intravaginal dehydroepiandrosterone (DHEA) on moderate to severe dyspareunia and vaginal dryness, symptoms of vulvovaginal atrophy, and of the genitourinary syndrome of menopause. Menopause. 2016 Mar;23(3):243-56. doi: 10.1097/GME.0000000000000571. PMID 26731686